CLINICAL TRIAL: NCT05463250
Title: Smartwatch and Physician Well-being: Are Wearables Part of the Solution?
Brief Title: Smartwatch and Physician Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Physicians Foundation (Unknown); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 22-0799
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Professional Burnout
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Smart Watch, then no intervention (Experimental): Physicians will be asked to wear a Smartwatch for 6 months, and then will be monitored for the following 6 months without wearing a Smartwatch. Physicians will complete surveys about their experiences
  Interventions: Device: Smartwatch
- No intervention, then Smart Watch (Experimental): Physicians will be monitored for the first 6 months without wearing a Smartwatch, and then will be asked to wear a Smartwatch for the following 6 months. Physicians will complete surveys about their experiences
  Interventions: Device: Smartwatch

INTERVENTIONS:
Device: Smartwatch — Wearing a smartwatch and having access to its data

SUMMARY:
The prevalence of burnout and other forms of distress among physicians is alarmingly high. This clinical trial is being conducted to learn more about if wearing a Smartwatch and having access to its data improves physicians' sense of well-being and if data measured from Smartwatches contain a 'signal' that predicts well-being

DETAILED DESCRIPTION:
We will conduct a randomized controlled trail to evaluate if wearing a Smartwatch improves overall well-being among physicians, and if so, in which dimension of well-being (e.g., fatigue, stress, overall quality of life, burnout). Additionally, we will explore if data from Smartwatches can predict subsequent well-being among physicians.

Study Aims:

1. To determine if wearing a Smartwatch and having access to its physiological data (e.g., sleep, step count, activity, breathing reminders) improves well-being, and if so which well-being dimensions.
2. To determine whether continuous physiological measures (measured from Smartwatches) contain a 'signal' that predicts physician well-being, and if so in which dimensions.

ELIGIBILITY:
Inclusion Criteria:

* Physician

Exclusion Criteria:

* non physicians

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Burnout | Up to 12 months
  The Maslach Burnout Inventory measures emotional exhaustion, depersonalization, and low sense of personal accomplishment. Possible scores range from 0-27 (emotional exhaustion subscale), 0-10 (depersonalization subscale), and 0-40 (personal accomplishment subscale). Higher scores on the emotional exhaustion and depersonalization subscales and lower scores on the personal accomplishment subscale indicates worse outcome.

SECONDARY OUTCOMES:
Physician Well-Being Index | Up to 12 months
  The Physician Well-Being Index measures multiple dimensions of distress (burnout, fatigue, quality of life, stress) and satisfaction with work-life integration and meaning in work. The total score ranges from -2 to 9, with higher scores indicating a greater degree of distress, lower meaning in work, and less satisfaction with work-life integration.

CONTACTS AND LOCATIONS:
Overall Officials: Liselotte N Dyrbye, MD MHPE, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- Lotte Dyrbye, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dyrbye LN, West CP, Wilton AR, Satele DV, Athreya AP. Smartwatch Use and Physician Well-Being: A Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2527275. doi: 10.1001/jamanetworkopen.2025.27275. PMID 40824640